CLINICAL TRIAL: NCT06599918
Title: Randomized, Double-blind, Placebo-controlled Study of the Efficacy and Safety of Nicotinamide in Patients With and Liver Fibrosis (NICOFIB)
Brief Title: Study of the Efficacy and Safety of Nicotinamide in Patients With Liver Fibrosis (NICOFIB)
Acronym: NICOFIB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIBSP-NIC-2021-157; 2023-504100-28 (EudraCT Number)
Record Dates: First submitted 2024-07-11; First posted 2024-09-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Fatty Liver; Obesity; Hepatic Fibrosis; NAFLD; Nicotinamide; Overweight and Obese Adults
Keywords: Nicotinamide; Fatty liver; Nafld
MeSH Terms: conditions — Fatty Liver; Obesity; Liver Cirrhosis; Non-alcoholic Fatty Liver Disease; Overweight | interventions — Niacinamide

STUDY DESIGN:
Intervention Model Description: A controlled, randomized, double-blind, and multicenter clinical trial has been designed to explore the proof-of-concept regarding the effects of nicotinamide (NAM) administration on hepatic inflammation and fibrosis in individuals with a BMI over 27. The trial adopts a parallel design, incorporating a placebo control group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will be double-blind. The delivery of the investigational product will not contain information about the assigned treatment arm or the administered dose. Both interventions will have the same presentation format and identical visual characteristics. Therefore, both the patient and the Endocrinology specialist facilitating the intervention will be unaware of the assigned treatment arm.
  All personnel from the sponsor and investigator's center involved in the study will undergo masking concerning the assigned treatment, with the following exceptions:
  The pharmacy staff at the center involved in the preparation. The Pharmacy Service at Sant Pau Hospital will mask the study medication, labeling it with consecutive code numbers following the randomization table.
  The sponsor's pharmacovigilance personnel reporting adverse events to health authorities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Administration of the placebo compound, in the same format as the active compound.
  The placebo is composed by microcrystalline Cellulose (Excipient No. 1 for capsules: 98.05% microcrystalline cellulose, 1.95% colloidal silica). Molecular formula: C14H26O11 IUPAC name: methyl 4-O-methyl-hexopyranosyl-(1->4)-hexopyranoside Molecular weight: 370.35 g/mol Qualitative and quantitative composition (per capsule): Microcrystalline Cellulose 400 mg Pharmaceutical form: Hard gelatin capsules containing. Dose and route of administration: maximum 2.4 g daily/oral. Raw material suppliers: Fagron and Acofarma. Encapsulation location: Pharmacy Service of HSCSP.
  Interventions: Drug: Placebo
- Nicotinamide (Active Comparator): Administration of the active compound, the amide form of vitamin B3, Nicotinamide (NAM).
  International Nonproprietary Name: Nicotinamide. Molecular formula: C6H6N2O IUPAC name: Pyridine-3-carboxamide. Molecular weight: 122.12 g/mol. Qualitative and quantitative composition (per capsule): Nicotinamide 500 mg. Pharmaceutical form: Hard gelatin capsules. Dose and route of administration: maximum 3 g daily/oral. Raw material suppliers: Fagron and Acofarma. Encapsulation location: Pharmacy Service of HSCSP.
  Interventions: Drug: Nicotinamide

INTERVENTIONS:
Drug: Nicotinamide — Administration of NAM on a variable dose depending on the participant's body weight. Administration is done orally, daily.
  Other Names: NAM
  Arms: Nicotinamide
Drug: Placebo — Administration of placebo on a variable dose depending on the participant's body weight. Administration is done orally, daily.
  Arms: Placebo

SUMMARY:
The objective of this clinical trial, a pilot study, is to assess the impact of nicotinamide (NAM) on individuals with hepatic fibrosis.

The main question it aims to answer is:

- To determine if the treatment with NAM is able to arrest, or even reduce, the hepatic fibrosis.

In addition, we also want to study the effect of NAM on:

* General parameters (weight, HOMA-IR, etc).
* Adiposity distribution (liver and body).
* Systemic inflammation.
* Thermogenic capacity of adipose tissue.
* Microbiota composition.

Researchers will compare NAM to a placebo, to see if NAM can arrest or revert hepatic fibrosis and its associated effects.

Participants will take either NAM or placebo. The dosage will be 1.2g/m2 NAM per day, for one year.

DETAILED DESCRIPTION:
Patients with a Fibroscan > 8 kPa will be offered to participate in this study. Participants will receive either placebo or a NAM dose adjusted to body weight. The duration of the treatment is 12 months.

Participants will be subjected to a total of 5 follow-up and/or control visits:

Visit 1

* Physical examination(weight, height, BMI, waist circumference, neck circumference, blood pressure, and heart rate).
* Assessment of muscle status and risk of sarcopenia: grip strength, chair test.
* Basal electrocardiogram.
* Blood analysis.
* Bioelectrical impedance analysis.
* Nuclear magnetic resonance.
* Thermographic image.
* Food questionnaire (PREDIMED).
* International Physical Activity Questionnaire (IPAQ).
* Collection of blood, urine, and feces samples for storage in the biobank.

Visit 2. Control visit (time month 1)

* Monitoring of adverse events (AE) and adverse reactions (AR).
* Electrocardiogram.
* Control blood analysis: sodium, potassium, liver biochemistry (AST, ALT, bilirubin, GGT, FA), renal function (urea, creatinine, estimated glomerular filtration), and coagulation tests.
* Physical examination and measurement of vital signs.

Visit 3. Follow-up visit (time month 3)

* Monitoring of AE and AR.
* Drug adherence questionnaire.
* Electrocardiogram.
* Blood analysis.
* Physical examination (weight, BMI, waist circumference, neck circumference, blood pressure, and heart rate).
* Collection of blood, urine, and feces samples for biobank.
* Collection of concomitant medication.
* Adherence to study treatment and dietary recommendations.

Visit 4. Follow-up visit (time month 6)

* Monitoring of AE and AR.
* Drug adherence questionnaire.
* Electrocardiogram.
* Blood analysis.
* Physical examination (weight, BMI, waist circumference, neck circumference, blood pressure, and heart rate).
* Collection of blood, urine, and feces samples for biobank.
* Collection of concomitant medication.
* Adherence to study treatment and dietary recommendations.

Visit 5. Control visit (time month 9).

* Monitoring of AE and AR.
* Drug adherence questionnaire.
* Electrocardiogram.
* Control blood analysis.
* Physical examination.
* Collection of concomitant medication.

Visit 6. Final exploration (time month 12)

* Monitoring of AE and AR.
* Drug adherence questionnaire.
* Food questionnaire (PREDIMED).
* Physical Activity Questionnaire (IPAQ).
* Physical examination and measurement of vital signs (weight, BMI, waist circumference, neck circumference, blood pressure, and heart rate).
* Assessment of muscle status and risk of sarcopenia: FPM, chair test.
* Electrocardiogram.
* Blood analysis.
* Measurement of NAM and derived metabolites in serum and urine.
* Nuclear magnetic resonance.
* Bioimpedance.
* Thermographic image.
* Fibroscan® with CAP.
* Collection of blood, urine, and feces samples for biobank

The safety of the participants will be assessed using a record of the AEs and ARs that could arise and their annotation in the EDC, as well as a regular evaluation of liver, kidney, and heart function at baseline, 1, 3, 6, 9 and 12 months

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 85 years.
* Diagnosis of non-alcoholic fatty liver disease (NAFLD) by their referring physicians (NAFLD defined as the presence of hepatic steatosis and in the absence of significant alcohol consumption, having excluded other liver diseases).
* BMI between 27-40 kg/m2.
* Fibroscan® value greater than 9.2 kPa, obtained within the last 6 months prior to the start of the study.

Exclusion Criteria:

* Patients with any medical condition or illness that, in the opinion of the investigator, could interfere with the study results and/or affect the patients' ability to participate or complete the study.
* History of clinically significant heart disease (ejection fraction <40% [normal range 50-70%], heart failure defined as New York Heart Association [NYHA] Class > 2; clinically significant congenital or acquired valvular disease; symptomatic coronary artery disease such as myocardial infarction or angina, history of unstable arrhythmias, history of atrial fibrillation).
* Decreased renal function (estimated glomerular filtration rate <45 mL/min/1.73 m2, calculated using the CKD-EPI formula) at screening.
* Alcohol consumption exceeding 30 g/day in men or 20 g/day in women.
* Patients with significant impairment of liver function in the selection analysis defined as repeated values of AST, ALT, and bilirubin > 3 times the upper limit of normal.
* Positive for hepatitis B surface antigen or hepatitis C antibodies.
* Patients with hepatocellular carcinoma.
* Patients with liver cirrhosis (Fibroscan® > 18, compatible biopsy, or those who have experienced decompensations of cirrhosis).
* Patients diagnosed with human immunodeficiency virus (HIV).
* Patients with hypersensitivity or a history of severe allergies to NAM or excipients used in the preparation of capsules (NAM and placebo).
* Patients with iodinated contrast allergy.
* History or evidence of an autoimmune disorder considered clinically significant by the investigator or requiring systemic, chronic use of systemic corticosteroids or other immunosuppressants.
* Patients on treatment with hepatotoxic drugs (amiodarone, immunosuppressants, ART, antituberculosis drugs, corticosteroids, etc.).
* Patients consuming narcotic and psychotropic substances with hepatotoxic effects.
* Individuals with incapacitating diseases or cognitive impairment.
* Institutionalized patients or those without a fixed address.
* Principal investigator's discretion in case of indications of low adherence to the trial or follow-up visits.
* Individuals with a life expectancy of less than 12 months.
* Patients participating in another interventional clinical trial, excluding observational/natural history studies, at the start of the study or within the last 30 days before the start of the study.
* Previous use of vitamin B3 (NAM), with abstinence required for at least 3 months before screening.
* Pregnant women as determined by a positive high-sensitivity serum or urine pregnancy test (minimum sensitivity of 25 IU/L or equivalent units of hCG) within 24 hours prior to screening, dosing, or completion of the study. Women of childbearing potential (WOCBP) will undergo a pregnancy test (serum or urine) 24 hours prior to screening, dosing, or completion of the study. Such participants must use a highly effective contraceptive method, such as combined hormonal contraceptives or intrauterine device (IUD), in accordance with the Clinical Trial Facilitation Group, throughout the entire study.
* Breastfeeding women.
* Patients undergoing treatment/supplementation with vitamin E.
* Patients receiving probiotics.
* Patients on the waiting list for bariatric surgery in the next 12 months.
* Patients undergoing treatment with drugs that may have an effect on the progression of liver disease.
* Drugs for the treatment of T2DM with effects on NAFLD (GLP-1 analogs, thiazolidinediones such as pioglitazone) initiated within 6 months before the study start.
* Drugs for the treatment of T2DM with effects on intestinal microbiota (metformin, α-GI inhibitors, DPP-4 inhibitors, and SGLT-2 inhibitors) initiated within 6 months before the study start.
* Patients who do not sign the informed consent.
* Patients with contraindications to the contrast agent to be used in imaging tests.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Effect of nicotinamide on hepatic fibrosis | Fibroscan at 0 and 12 months.
  Measurement of hepatic fibrosis by Fibroscan, to asses the arrest or improvement of fibrosis (lower value than basal Fibroscan result)

SECONDARY OUTCOMES:
Effect of nicotinamide on body fat and hepatic fat distribution | 0 and 12 months
  Analysis of body and hepatic fat by magnetic ressonance and observe visual differences between the basal and final images
Effect of nicotinamide on the general health state (weight) | Blood test and strength test at 0, 3, 6, and 12 months
  Analysis of body weight (grams) and waist circumference (cm), a reduction in both would point to a better general status and a weight loss
Effect of nicotinamide on the general health state (strenght) | Blood test and strength test at 0, 3, 6, and 12 months
  Evaluation of the grip strength as a measure of muscle strength
Effect of nicotinamide on the Insulin resistance | Blood test and strength test at 0, 3, 6, and 12 months
  Calcutaltion of the HOMA-IR (homeostatic model assessment - Insulin Resistance) index, a reduction of the HOMA-IR index shows a reduction of insulin resistance and an improved glucose metabolism
Effect of nicotinamide on gut microbiota | Test at 0, 3, 6, and 12 months
  Analyses of the gut microbiota composition during the NAM treatment
Effect of nicotinamide on systemic inflammation | Blood test at 0, 3, 6, and 12 months
  Analysis of the evolution of systemic inflammation by ELISA (enzyme-linked immunosorbent assay) of several cytokines related to inflammation. Lower values are usually associated to lower inflammation.
Effect of nicotinamide on cellular inflammation | Blood test at 0, 3, 6, and 12 months
  Analysis of the evolution of cellular inflammation by analyzing the count and type of peripheral blood mononuclear cells by flow-cytometry
Security evaluation LIVER | 0, 1, 3, 6, 9, and 12 months
  Security evaluation of the dosage of nicotinamide administered by analyzing liver parameters of aspartate transaminase (AST), alanine transaminase (ALT), and coagulation parameters.
Security evaluation KIDNEY | 0, 1, 3, 6, 9, and 12 months
  Security evaluation of the dosage of nicotinamide administered by measuring glomerular filtrate and creatinine
Effect of nicotinamide on liver parameters | 0 and 12 months
  Evaluation of the effects of nicotinamide on liver status by ELF-test, to observe if there is any improvement (lower value than basal measurement)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided